CLINICAL TRIAL: NCT04748640
Title: Bilateral Essential Tremor Treatment With Gamma Knife
Acronym: BEST-GK
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Christian Iorio-Morin, Assistant professor of neurosurgery, Université de Sherbrooke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-5172
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Essential Tremor
Keywords: Gamma Knife Thalamotomy; Tremor; Essential Tremor; Dyskinesias; Neurologic Manifestations; Nervous System Diseases; Movement Disorders; Central Nervous System Diseases
MeSH Terms: conditions — Essential Tremor; Tremor; Dyskinesias; Neurologic Manifestations; Nervous System Diseases; Movement Disorders; Central Nervous System Diseases

STUDY DESIGN:
Masking Description: All assessments filmed on video and scored by a blinded evaluator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Participants will undergo a thalamotomy contralateral to their previous treatment with Gamma Knife using a frame-based, Gamma Knife Perfexion or Icon unit (Elekta, Stockholm, Sweden).
  Interventions: Procedure: Gamma Knife VIM thalamotomy

INTERVENTIONS:
Procedure: Gamma Knife VIM thalamotomy — Ablation of contralateral VIM nucleus of thalamus with GK using a frame-based, Gamma Knife Perfexion or Icon unit (Elekta, Stockholm, Sweden).

SUMMARY:
Combined Phase II/III, multi-center, prospective, single-blinded trial.

Ten (10) patients with essential tremor who previously underwent successful and uncomplicated GK thalamotomy for essential tremor will undergo a contralateral treatment. The incidence of side effects will be determined at 3 months postoperatively, graded per the CTCAE v5 and analyzed by a data safety monitoring board. Upon successful review, this Phase II trial will be converted to a Phase III trial of utility that will enrol 40 additional patients. The primary outcome will be the change in QUEST score at 12 months postoperatively, as well as a patient-reported assessment of Health Utility. Secondary outcomes will include objective tremor, gait and speech assessments (filmed and scored by blinded evaluators), as well as quality of life questionnaires and adverse events questionnaires. Outcomes will be assessed at baseline, as well as 3, 6, 12, 24 and 36 months post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 18 years
* The patient has a primary diagnosis of ET or ET plus confirmed by a movement disorder neurologist;
* The patient previously underwent a GK thalamotomy (> 12 months ago);
* The tremor on the untreated side negatively impacts the patients' quality of life;
* The patient wants treatment of the contralateral side.

Exclusion Criteria:

* Clinically relevant gait and/or balance impairment (e.g. wide-based, more than 2 falls/months, wheelchair, walker, cane use);
* Clinically relevant speech impairment (e.g. impairment of intelligibility);
* Inability to comply with the follow-up schedule;
* Refusal of the treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-06-08 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in QUEST Score | 12 months
  Difference in QUEST score between baseline and the 12-month follow-up, with statistical significance defined as p = 0.05 and a minimum clinically important difference (MCID) defined as 5
Patient-based Assessment of Utility | 12 months
  A patient-reported assessment of utility after 12 months using the question "Knowing what you know now, would you do this treatment again?".

SECONDARY OUTCOMES:
Gait Assessment (NRS-11) | Baseline, post operative month 3, 6, 12, 24, 36
  Patient-reported and blinded observer rating of the patient's ability to walk (Numerical rating scale (NRS-11) from 0 to 10, with 10 being best)
Gait Assessment (missteps) | Baseline, post operative month 3, 6, 12, 24, 36
  Number of missteps in a 6 m standardized tandem walk
Falls | Baseline, post operative month 3, 6, 12, 24, 36
  Number of falls in last month
Speech Assessment (NRS-11) | Baseline, post operative month 3, 6, 12, 24, 36
  Patient-reported and blinded observer rating of the patient's ability to speak (Numerical rating scale (NRS-11) from 0 to 10, with 10 being best)
Numbness | Baseline, post operative month 3, 6, 12, 24, 36
  Incidence of new-onset numbness
Dysgeusia | Baseline, post operative month 3, 6, 12, 24, 36
  Incidence of taste alterations
Other adverse events | Baseline, post operative month 3, 6, 12, 24, 36
  Incidence of other adverse events as classified in the CTCAE
Tremor (CRST) | Baseline, post operative month 3, 6, 12, 24, 36
  Assessment of tremor using the Clinical Rating Scale for Tremor (CRST) parts A (0-88) and B (0-36), higher scores correspond to a worse tremor).
Quality of life (QUEST) | Baseline, post operative month 3, 6, 12, 24, 36
  QUality of life in ESsential Tremor (QUEST) questionnaire (0-100 percent, higher scores correspond to a worse quality of life)
Quality of life (CRST part C) | Baseline, post operative month 3, 6, 12, 24, 36
  Part C of the Clinical Rating Scale for Tremor (CRST) (0-32, higher scores correspond to a worse quality of life)
Health Utility (EQ-5D-5L) | Baseline, post operative month 3, 6, 12, 24, 36
  Health Utility measured using the EQ-5D-5L and computed using the Canadian preference weights. Values range from 0 to 1, with 1 representing a perfect health.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Toronto Western Hospital, University Health Network, Toronto, Ontario
  - CIUSSS de l'Estrie-CHUS - Hôpital Fleurimont, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No